CLINICAL TRIAL: NCT01749631
Title: A Prospective, Open-label, Multicenter, Post Marketing, Observational Study to Investigate the Effectiveness of Sevoflurane Anaesthesia in Difficult to Intubate Egyptian Patients
Brief Title: Investigation of the Effectiveness of Sevoflurane Anaesthesia in Difficult to Intubate Egyptian Patients
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P13-805
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Intubation; Difficult
Keywords: Patients suspected to have difficult intubation; Intratracheal intubation; Difficult to intubate

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Difficult to Intubate (DTI) Participants: Male or non-pregnant females over 18 years of age with Mallampati score III or IV who were undergoing surgery using sevoflurane as the anesthetic agent as judged by the investigator and in compliance with the drug market authorization and approved product labeling.

SUMMARY:
The purpose of this study was to record the effectiveness of sevoflurane for intubation in Egyptian, non-obstetric, difficult to intubate (DTI) patients undergoing surgery in regards to the rate of intubation success.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicenter, post marketing, observational study to investigate the effectiveness of sevoflurane anaesthesia in difficult to intubate (DTI; Mallampati Score III or IV) Egyptian patients who had been prescribed sevoflurane for anaesthesia by their treating physician.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female over 18 years who are undergoing surgery and using sevoflurane as the anesthetic agent and with Mallampati score III or IV

2. Patients with at least one of the below criteria:

1. Anatomic

   * micrognathia - small mandible
   * macroglossia - large tongue
   * short or fixed neck
   * anterior vocal cords
2. Trauma - neck or face
3. Burns - airway edema
4. Infections - edema

   * Retropharyngeal abscess
   * Submandibular abscess
   * epiglottitis
   * laryngotracheobronchitis (croup)
5. Neoplasms; e.g., laryngeal tumors
6. Rheumatoid arthritis - temporomandibular joint (TMJ) immobility
7. Diabetes mellitus
8. Waxy skin - palm test
9. Decreased functional residual capacity (FRC) - rapid desaturation (due to displaced diaphragm, increased closing capacity and small airway closure, increased oxygen consumption)
10. airway closure in supine position
11. Morbid obesity (body mass index [BMI] >35)
12. Airway edema
13. Laryngospasm
14. Edentulous patients - indent cheeks.

3. Patients willing to sign informed consent

Exclusion Criteria:

1. Patients with present use of opioids and/or narcotic dependent.
2. Patients with known sensitivity to sevoflurane or to other halogenated agents.
3. Patients with known or suspected genetic susceptibility to malignant hyperthermia.
4. Alcohol addictive patients.
5. Patients with Renal insufficiency (baseline serum creatinine greater than 1.5 mg/dL)
6. Patient is a pregnant or breastfeeding female

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitals with operation theaters
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2012-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amr Alaa, Study Director — AbbVie Egypt

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 97 participants were enrolled and included in the intent-to-treat (ITT) population; 1 participant did not meet the criteria Mallampati Score III or IV and was excluded from the per protocol population, which consisted of 96 participants.
Period: Overall Study
Arm/Group | Difficult to Intubate (DTI) Participants
Started | 97
Completed | 97
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Per protocol population: all participants prescribed sevoflurane due to an anticipated difficulty in intubation during surgery and who met the study's inclusion/exclusion criteria.
Arm/Group | Difficult to Intubate (DTI) Participants
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (15.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Intubation (Clinical Success)
Description: Participants were considered to have a successful intubation if intubation was achieved in less than 4 separate intubation attempts according to the guidelines of the American Society of Anesthesiologists (ASA). The number of intubation attempts was a maximum of 3 attempts, after which the intubation was considered a failure.
Time Frame: Start of intubation to completion of intubation (up to 15 minutes)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Difficult to Intubate (DTI) Participants
Number analyzed (Participants) | 96
percentage of participants
  Success | 96.9
  Failure | 3.1

2. Secondary Outcome: Mean Duration of Induction (in Seconds)
Description: The mean duration of induction (in seconds) was defined as the time required to reach a Ramsay Sedation Score (RSS) of 5 from start of induction. The RSS levels are defined as 1 = anxious, agitated or restless; 2 = calm, co-operative and communicative; 3 = response is quick to a voice command; 4 = response is slow to a voice command; 5 = slow or sluggish response; and 6 = no response at all.
Time Frame: From start of induction up to 15 minutes
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Difficult to Intubate (DTI) Participants
Number analyzed (Participants) | 96
seconds | 220.45 (23.43)

3. Secondary Outcome: Percentage of Participants With Mallampati Score III and IV
Description: Mallampati classification correlates tongue size to pharyngeal size. The test is performed with the patient in the sitting position, head in a neutral position, the mouth wide open and the tongue protruding to its maximum, without phonation. Classification is assigned according to the extent the base of tongue is able to mask the visibility of pharyngeal structures: Class I = visualization of the soft palate, fauces; uvula, anterior and the posterior pillars; Class II = visualization of the soft palate, fauces and uvula; Class III = visualization of soft palate and base of uvula; and Class IV: only hard palate is visible, soft palate is not visible at all. A high score (Class III or IV) is associated with more difficult intubation.
Time Frame: Screening
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Difficult to Intubate (DTI) Participants
Number analyzed (Participants) | 96
percentage of participants
  Class III | 93.8
  Class IV | 5.2

4. Secondary Outcome: Mean Duration of Intubation Procedure (in Minutes)
Description: The mean duration of intubation procedure (in minutes) was defined as the time from intubation start to the completion of the intubation process (from tube introduction to partial pressure of end-tidal carbon dioxide [PETCO2]).
Time Frame: Start of intubation to completion of intubation (up to 15 minutes)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Difficult to Intubate (DTI) Participants
Number analyzed (Participants) | 96
minutes | 1.77 (0.2)

5. Secondary Outcome: Percentage of Participants Who Experienced Complications Resulting From Intubation Procedure
Description: The percentage of participants who experienced complications resulting from the intubation procedure including, but not limited to, bleeding, salivating, and lung aspiration.
Time Frame: Start of intubation to completion of intubation (up to 15 minutes)
Population: ITT population: all participants prescribed sevoflurane due to an anticipated difficulty in intubation during surgery.
Measure: Number; unit: percentage of participants
Arm/Group | Difficult to Intubate (DTI) Participants
Number analyzed (Participants) | 97
percentage of participants
  Hypertension | 1.03
  Cough | 1.03

6. Secondary Outcome: Percentage of Participants Who Experienced Difficulties Related to the Use of Sevoflurane
Description: The percentage of participants who experienced difficulties related to the use of sevoflurane including, but not limited to, vocal cords adduction, coughing, movements, and apnea episodes.
Time Frame: From start of induction to completion of intubation (up to 30 minutes)
Population: ITT population: all participants prescribed sevoflurane due to an anticipated difficulty in intubation during surgery.
Measure: Number; unit: percentage of participants
Arm/Group | Difficult to Intubate (DTI) Participants
Number analyzed (Participants) | 97
percentage of participants | 0

7. Secondary Outcome: Mean Number of Intubation Attempts
Time Frame: Start of intubation to completion of intubation (up to 15 minutes)
Population: as for baseline characteristics
Measure: Mean (Standard Error); unit: number of attempts
Arm/Group | Difficult to Intubate (DTI) Participants
Number analyzed (Participants) | 96
number of attempts | 1.26 (0.50)

ADVERSE EVENTS:
Time Frame: All AEs were collected from the time of study drug administration to end of intubation procedure (up to 30 minutes); SAEs were also collected from the time that informed consent was obtained until 30 days after last dose of study drug (30 days).
Arm/Group | Difficult to Intubate (DTI) Participants
Serious Adverse Events (participants affected / at risk) | 0/97
Other Adverse Events (participants affected / at risk) | 2/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Difficult to Intubate (DTI) Participants (N=97)
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.